CLINICAL TRIAL: NCT05905016
Title: Prospective Evaluation of the Clinical Utility of Peroral Endoscopic Myotomy for Gastrointestinal Motility Disorders
Acronym: POEM
Status: Recruiting | Type: Observational
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Other Study IDs: 1798543
Record Dates: First submitted 2022-02-23; First posted 2023-06-15 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Achalasia; Esophageal Spasm, Diffuse; Gastroparesis; Swallowing Disorder; Zenker Diverticulum
MeSH Terms: conditions — Esophageal Achalasia; Esophageal Spasm, Diffuse; Gastroparesis; Deglutition Disorders; Zenker Diverticulum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Esophageal POEM: Data will be collected for patients under going standard of care Esophageal POEM (E-POEM)
- Gastric POEM: Data will be collected for patients under going standard of care Gastric POEM (G-POEM)
- Zenker's POEM: Data will be collected for patients under going standard of care Zenker's diverticulum POEM (Z-POEM)

SUMMARY:
This is prospective data recording study. All patients will receive standard medical care and no experimental interventions will be performed.

DETAILED DESCRIPTION:
This is prospective data recording study. All patients will receive standard medical care and no experimental interventions will be performed.

This study will enroll 600 subjects over the next 4 to 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. Scheduled to undergo POEM

Exclusion Criteria:

1. Any contraindication to performing endoscopy.
2. Participation in another research protocol that could interfere or influence the outcomes measures of the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who present to the Center for Interventional Endoscopy for standard of care POEM procedures.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Post procedural Reflux Rate | 12 months
  Rate of Long-Term Clinical Success and Post-procedural Reflux Rate Among Patients with Esophageal Dysmotility Undergoing POEM
Long-Term Clinical Efficacy of G-POEM for the management of medically refractory gastroparesis | 12 months
  The main outcome of the study is to evaluate the proportion of patients who have clinical response to GPOEM. Clinical response is measured by the validated symptom assessment tool (gastroparesis cardinal symptom index - GCSI). Patients with a decrease in GCSI by one or more point will be defined as having a clinical response.
Long-Term Clinical Efficacy of Z-POEM for the management of Zenker's Diverticulum and Rate of Recurrence | 12 months
  The main outcome of this study is to evaluate rate of recurrence of symptoms after Z-POEM for Zenker's diverticulum. Recurrence is defined as a return of patient's symptoms (dysphagia, odynophagia) at the time of clinic follow-up.
Evaluate the efficacy of POEM for the management of gastrointestinal disease for esophageal motility. | 12 months
  The main outcome measure is to evaluate the long-term efficacy of POEM for esophageal motility disorders. Efficacy or clinical response is usually assessed using the Eckardt score. An Eckardt score of < 3 is traditionally defined as treatment response following POEM.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Yang, MD, Principal Investigator — AdventHealth Orlando
Locations (1):
- AdventHealth Orlando, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No